CLINICAL TRIAL: NCT01811823
Title: Effect of HIV and/or Active Tuberculosis on the Humoral and Cell Mediated Immune Responses to Un-adjuvanted Trivalent Sub-unit Influenza Vaccine (TIV) in Adults
Brief Title: Effect of HIV and/or Active Tuberculosis on the Immune Responses to Trivalent Influenza Vaccine (TIV) in Adults
Acronym: TIV_HIV_TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Shabir Madhi, Dr, University of Witwatersrand, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TIV_HIV_TB
Record Dates: First submitted 2013-02-21; First posted 2013-03-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Influenza; HIV; Tuberculosis
Keywords: Tuberculosis; HIV infection; Immune responses to Influenza vaccination
MeSH Terms: conditions — Influenza, Human; Tuberculosis; HIV Infections | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TIV (Other): Trivalent Inactivated Influenza Vaccine The study vaccine will be the seasonal 2013 un-adjuvanted TIV which is provided as a 0•5 milliliter suspension of split virus mixture of 15 micrograms each of circulating H1N1- like strain, H3N2- like strain and B - like strain.
  The WHO recommended vaccine formulation for Southern Hemisphere 2013 Influenza Season contains the following influenza strains:
  * A/California/7/2009 (H1N1)pdm-like virus
  * A/Victoria/361/2011 (H3N2)-like virus
  * B/Wisconsin/1/2010-like virus. (Yamagata lineage)
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza Vaccine — The study vaccine will be the seasonal 2013 un-adjuvanted TIV which is provided as a 0•5 milliliter suspension of split virus mixture of 15 micrograms each of circulating H1N1- like strain, H3N2- like strain and B - like strain.
  The WHO recommended vaccine formulation for Southern Hemisphere 2013 Influenza Season contains the following influenza strains:
  * A/California/7/2009 (H1N1)pdm-like virus
  * A/Victoria/361/2011 (H3N2)-like virus
  * B/Wisconsin/1/2010-like virus. (Yamagata lineage)
  Other Names: Vaxigrip

SUMMARY:
Prospective, open-labelled study which will enrol 360 participants in four groups of 80 participants including: HIV-uninfected adults without evidence of TB; HIV-infected adults without any evidence of TB; HIV-uninfected adults with concurrent microbiologic confirmed TB, HIV-infected adults with concurrent microbiologic confirmed TB.

Participants will receive the recommended seasonal 2013 un-adjuvanted Trivalent Influenza Vaccine (TIV). At 3 visits, blood will be collected for determination of immune responses.

Objective:

• To determine the effect of HIV-infection, tuberculosis (TB) and HIV-TB co-infection on immune responses

ELIGIBILITY:
Inclusion Criteria:

* for HIV-infected subjects: a Cluster of Differntiation4 (CD4+) cell count of >100/ul within the previous 3 months;
* able to attend the clinic for immunogenicity and illness visits;
* for subjects with TB: having a microbiologic confirmed diagnosis of TB (defined as the presence of acid-fast-bacilli (AFB) on a sputum smear or other specimen and/or a positive culture for M. tuberculosis) within the past 120 days;
* Aged 18 to 55 years.

Exclusion Criteria:

* any contraindication to influenza vaccine;
* any contraindication to intramuscular injections;
* any existing grade 3 or grade 4 laboratory or clinical toxicity as per Division of Acquired Immune Deficiency Syndrome (DAIDS) toxicity tables;
* systemic steroid treatment for >21 days within the past 30 days.
* pregnancy (a urine Human Chorionic Gonadotropin (βHCG) will be performed on all women of childbearing age to exclude pregnancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2014-11-20 (Actual)

PRIMARY OUTCOMES:
humoral antibody responses, measured by hemagglutinin inhibition assay (HAI), to each of three strains included in the seasonal non-adjuvanted trivalent influenza vaccine. | up to 6 weeks after end of the influenza season
  • To determine the effect of HIV-infection, tuberculosis (TB) and HIV-TB co-infection on humoral antibody responses, measured by hemagglutinin inhibition assay (HAI), to each of three strains included in the seasonal non-adjuvanted trivalent influenza vaccine In this study we will use the following definitions to assess the humoral immune response to TIV: HAI titers <1:10 = seronegative; HAI titers ≥1:10 = seropositive; HAI titers ≥1:40 = sero-protective; sero-response rate (primary outcome measure) will be defined as a titer of ≥1:40 in an individual with baseline titers of <1:10, or >4-fold increase of HAI titers if baseline titers were ≥1:10. Hemagglutination inhibition assays will be performed on serum as per recommended methods. Sera will be titrated against antigens from the influenza vaccine strains included in the 2013 seasonal TIV.

SECONDARY OUTCOMES:
• To compare the effect of HIV-infection, tuberculosis (TB) and HIV-TB co-infection on vaccine-strain specific cell mediated immune responses, evaluated by ELISPOT assay, following non-adjuvanted TIV vaccination. | up to 6 weeks after the end of the influenza season
  • To compare the effect of HIV-infection, tuberculosis (TB) and HIV-TB co-infection on vaccine-strain specific cell mediated immune responses, evaluated by Enzyme-linked immunosorbent spot (ELISPOT) assay, following non-adjuvanted TIV vaccination.
  The cell mediated Immunity (CMI) evaluations in this study will provide novel information on influenza-specific CMI in individuals with TB. Interferon gama- ELISPOT responses will be assessed on fresh Peripheral Blood Mononuclear Cells (PBMCs). Spots will be visualized with a ELISPOT plate reader. Background (non-specific) spots detected in the medium-containing wells will be subtracted from the wells stimulated with influenza antigens. Results will be reported as Spot forming cell (SFC)/106 PBMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, PHD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Respiratory and Meningeal Pathogens research unit, Johannesburg, Gauteng, South Africa